CLINICAL TRIAL: NCT00948623
Title: Physical Activity Counseling During Pulmonary Rehabilitation: Does it Improve Daily Physical Activity Levels
Brief Title: Physical Activity Counseling During Pulmonary Rehabilitation
Acronym: PAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Prof. Dr. T. Troosters, Department of Rehabilitation Sciences, Catholic University Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: s06081980
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; physical activity; pulmonary rehabilitation; counseling
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: physical activity counseling program
- 2 (Sham Comparator)
  Interventions: Behavioral: sham counseling program

INTERVENTIONS:
Behavioral: physical activity counseling program
  Arms: 1
Behavioral: sham counseling program
  Arms: 2

SUMMARY:
This randomized controlled trial will assess the effect of adding intensive physical activity counseling to an outpatient pulmonary rehabilitation program. Counseling including real-time feedback on daily activities from an activity monitor will be offered to improve participation in physical activities in daily life during and after an outpatient pulmonary rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Spirometry-proven COPD
* Referred for 6-month outpatient pulmonary rehabilitation program

Exclusion Criteria:

* Orthopedic problems impairing daily activities
* Progressive neurological or neuromuscular disorders
* Psychiatric or cognitive disorders
* Patients on the waiting list for lung transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Walking time in daily life and the amount of time spent in moderate intense activities

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Sciences, University Hospitals KULeuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Burtin C, Langer D, van Remoortel H, Demeyer H, Gosselink R, Decramer M, Dobbels F, Janssens W, Troosters T. Physical Activity Counselling during Pulmonary Rehabilitation in Patients with COPD: A Randomised Controlled Trial. PLoS One. 2015 Dec 23;10(12):e0144989. doi: 10.1371/journal.pone.0144989. eCollection 2015. PMID 26697853
- [Derived] Demeyer H, Burtin C, Van Remoortel H, Hornikx M, Langer D, Decramer M, Gosselink R, Janssens W, Troosters T. Standardizing the analysis of physical activity in patients with COPD following a pulmonary rehabilitation program. Chest. 2014 Aug;146(2):318-327. doi: 10.1378/chest.13-1968. PMID 24603844